CLINICAL TRIAL: NCT01747304
Title: Evaluation of Dual Energy X-ray Absorptiometry Scanners in the Identification of Atypical Femur Fractures - A Validation Study
Brief Title: Evaluation of IVA (SE Femur Scans) to Identify Incomplete AFFs
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 12-0352
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Atypical Femur Fracture
Keywords: Atypical Femur Fracture; DXA

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Screening population: Healthy post-menopausal women attending bone mineral density screening clinic with leg/hip/groin pain/discomfort/weakness an has been on anti-resorptive therapy for at least 5 years.
  Interventions: Device: DXA Se femur scans (previously called IVA femur)
- Comparator Group: Control group from Toronto CaMOS cohort willing to participate.
  Interventions: Device: DXA Se femur scans (previously called IVA femur)
- AFF group: participants in the AFF Cohort study at UHN
  Interventions: Device: DXA Se femur scans (previously called IVA femur)

INTERVENTIONS:
Device: DXA Se femur scans (previously called IVA femur) — Single Energy Beam (previously called inter-vertebral assessment) by Dual energy x-ray absorptiometry of affected femur
  Other Names: SF Femur scans

SUMMARY:
DXA scanners are routinely used to assess bone mineral density (BMD) and fracture risk in osteoporosis patients. They provide detailed bone imaging in a low radiation setting. Hologic manufactures scanners that are able to perform high definition instant vertebral fracture assessment (HD-IVA) used to screen at-risk patients for asymptomatic spine fractures instantly and reliably at the same time they are having their yearly BMD. We wish to investigate whether this same proven technology (HD-IVA scan mode) used on femurs (the scan mode is now called SE Femur scans) can be used to screen for atypical fractures of the femur in patients at risk for these debilitating fractures. In this proof of concept study, we propose to examine whether DXA scanners can provide a sensitive low radiation screening method to identify incomplete AFFs in patients with known incomplete AFFs and in patients at risk.

ELIGIBILITY:
Inclusion Criteria:

Known AFF group

1. A subject must have experienced an incomplete atypical low trauma fracture of the femoral shaft;
2. Is a patient at the UHN osteoporosis clinic.

Comparison Group

1. Must be scheduled for a bone mineral density scan at UHN
2. Have been on any bisphosphonate for 5 years or longer, and;
3. Have unexplained symptoms of leg, hip, thigh, or knee pain.

Exclusion Criteria:

* There are no exclusions

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Osteoporosis/Bone Mineral Density Lab out-patients
Sampling Method: Non-Probability Sample
Enrollment: 285 (Actual)
Dates: Start 2012-07; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
HD-IVA visualization of incomplete femur fractures | 1 day (one time point )
  Hologic DXA scanner using the high-definition IVA (HD-IVA) mode on femur bones will be able to visualize incomplete femur fractures at least 90% of the time in patients with known incomplete AFF.

CONTACTS AND LOCATIONS:
Overall Officials: Angela M Cheung, MD, PhD, CCD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada